CLINICAL TRIAL: NCT07131761
Title: Effect of Tai Chi Versus Moderate-intensity Combined Exercise Training on Cardiovascular Health and Physical Functional Performance in Older Men and Women With T2DM
Brief Title: Effect of Tai Chi Versus Moderate-intensity Combined Exercise Training on Cardiovascular Health and Physical Functional Performance in Older Men and Women With T2DM: the Tai Chi Intervention for Diabetes Management During Aging (TIDA) Study
Acronym: TIDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Emmanuel Gomes Ciolac, Full Professor of Department of Physical Education, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7.645.757
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes; Type 2 Diabetes; Cardiovascular risk factor; Metabolic risk; Non communicable disease; Vascular aging
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Noncommunicable Diseases | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi (Experimental): 40-60 minute supervised Yang-style Tai Chi lesson (24-form simplified pattern). Focus on calm, controlled movements and breathing coordination.
  Interventions: Other: Tai chi
- Moderate-Intensity Exercise (MICE) (Experimental): The MICE session will consist of five minutes of warm-up (joint mobility and stretching exercises between PSE levels 9 and 11, 30 minutes of walking on the treadmill between PSE levels 12 and 13, 20 minutes of muscle strengthening exercises between levels 12 and 14 of PSE (two sets of 15 to 20 repetitions in circuit in the exercises bent row with elastic band, bodyweight squats, adapted push-ups (on the wall or on the counter), deadlifts with an elastic band, presses with an elastic band and an abdominal band on the floor or adapted on the chair) and five minutes of back to calm (light stretching and breathing exercises at PSE level 9).
  Interventions: Other: Moderate-Intensity Combined Exercise (MICE)
- Control (No Exercise) (Experimental): The CON session will consist of 60 minutes of rest in the sitting position. Participants will be told not to sleep and will not have access to reading or electronic devices during the CON session.
  Interventions: Other: Control ( No Exercise )

INTERVENTIONS:
Other: Tai chi — Yang style of Tai Chi (24 form)
  Other Names: Tai Ji; Tai Chi Chuan
  Arms: Tai Chi
Other: Moderate-Intensity Combined Exercise (MICE) — start from warm up (5 minute )repetitions in circuit in the exercises bent row with elastic band, bodyweight squats, adapted push-ups (on the wall or on the counter), deadlifts with an elastic band, presses with an elastic band and an abdominal band on the floor or adapted on the chair and cool down in the end
  Arms: Moderate-Intensity Exercise (MICE)
Other: Control ( No Exercise ) — The CON session will last 60 minutes and will be conducted only sitting. Participants will be told not to sleep and will not be allowed to use reading materials or any electrical gadgets during the CON session.
  Arms: Control (No Exercise)

SUMMARY:
This randomized, single-blind, controlled clinical trial compares the effects of a 12-week Tai Chi program versus moderate-intensity combined exercise (MICE) training on cardiovascular health, glycemic control, and physical function in older adults with type 2 diabetes (T2DM). Sixty-six participants (33 men and 33 women) will be randomized 1:1:1 to Tai Chi (n = 22), MICE (n = 22), or a non-exercise control group (CON, n = 22).

The Tai Chi intervention involves three weekly Yang-style sessions, progressively increasing in duration and complexity while maintaining perceived exertion (PSE) below 12 (6-20 scale). The MICE program combines moderate-intensity walking (PSE 12-13) with six strengthening exercises (PSE 12-14), gradually increasing from 15 to 30 minutes/session and 1 to 3 sets over 12 weeks.

Primary outcomes include cardiovascular health (Life's Essential 8 index: diet, physical activity, nicotine exposure, sleep, BMI, lipids, blood glucose, and blood pressure) and glycemic control (fasting glucose, HbA1c). Secondary outcomes assess physiological mechanisms (heart rate variability, pulse wave velocity, flow-mediated dilation, carotid intima-media thickness), physical performance (6-minute walk test, grip strength, timed up-and-go), and quality of life (WHOQOL-BREF/OLD).

All evaluations will be conducted by blinded assessors under standardized conditions (21-24°C, morning fasting), except the 6MWT. Statistical analysis includes intention-to-treat repeated-measures ANOVA, ANCOVA for baseline adjustments, and per-protocol/adherence-adjusted analyses. Sample size (GPower) was calculated to detect a 0.8% HbA1c reduction with 90% power (30% attrition accounted for). An interim analysis at 50% completion will evaluate effect sizes/variability, with potential sample-size recalibration by an independent committee.

The study employs rigorous quality controls: standardized protocols, blinded assessments, and monitoring of confounders (medication changes, acute exercise effects). Ethical approval (CAAE: 88582225.1.0000.5398) ensures adherence to informed consent and privacy. By determining whether Tai Chi offers comparable or superior benefits to MICE for cardio metabolic health and functional capacity, this trial aims to inform evidence-based exercise prescriptions for older T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

only with type 2 diabetes

Exclusion Criteria:

* if not able to perform physical exercise (Extreme neuropathy, wounds in the feet, and amputation risk.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Health Score | At baseline (week 0) and after follow-up (week 12)
  Life's Essential 8 Index (0-100 scale)
  Components:
  Health behaviors: Diet, physical activity, nicotine exposure, sleep quality Health factors: BMI, blood lipids, blood glucose, blood pressure
Fasting Plasma Glucose | At baseline (week 0) and after follow-up (week 12)
  Change in fasting plasma glucose (FPG) levels (measured in mg/dL).
Glycated Hemoglobin (HbA1c) | baseline (Week 0) to follow-up (Week 12).
  Change in glycated hemoglobin (HbA1c) levels (measured as % of total hemoglobin)

SECONDARY OUTCOMES:
Carotid-femoral pulse wave velocity (PWVcf) | At baseline (week 0) and after follow-up (week 12)
  Carotid-femoral pulse wave velocity (PWVcf) will be measured using an automated device (Complior Analyze™ PWV and Central Pressure Analysis™; AlamMedical, Saint-Quentin-Fallavier, France), in meters per second (m/s)
Brachial artery flow-mediated dilation (FMD) | At baseline (week 0) and after follow-up (week 12)
  Change in brachial artery flow-mediated dilation (FMD) (%), calculated as:
  (peak diameter - baseline diameter) / baseline diameter × 100, measured via ultrasound (SonoSite M-Turbo™) after 5-minute artery occlusion.
Carotid Intima-Media Thickness | At baseline (week 0) and after follow-up (week 12)
  CIMT will be quantified using high-resolution B-mode ultrasound (SonoSite M-Turbo®, Fujifilm Inc., USA) with a 6-13 MHz linear array transducer with participants in the supine position and head rotated 45° contralaterally.
Central blood pressures | At baseline (week 0) and after follow-up (week 12)
  Central blood pressures will be assessed directly from the carotid pressure waveform, in millimeters of mercury (mmHg), and using a non-invasive automated device (Complior Analyze™ PWV and Central Pressure Analysis™; AlamMedical, Saint-Quentin-Fallavier, France)
Brachial blood pressure (BP) | At baseline (week 0) and after follow-up (week 12)
  Systolic and diastolic brachial blood pressure (BP) will be measured using an automatic monitor (Omron HEM 7200™, Omron Healthcare Inc., Dalian, China) in millimeters of mercury (mmHg)
Heart rate variability (HRV) - frequency domain | At baseline (week 0) and after follow-up (week 12)
  Frequency domain of heart rate variability (HRV) will be assesseded using a digital telemetry system (Polar H10™, Polar Electro Inc, Kempele, Finland) to measure HR signals beat-to-beat. A sequence of 256 stable R-R intervals will be used to calculate frequency in hertz (Hz).
Heart rate variability (HRV) - time domain | from baseline (Week 0) to follow-up (Week 12)
  Time domain of heart rate variability (HRV) will be assesseded using a digital telemetry system (Polar H10™, Polar Electro Inc, Kempele, Finland) to measure HR signals beat-to-beat. A sequence of 256 stable R-R intervals will be used to calculate time domain in milliseconds (ms).
Endurance performance | At baseline (week 0) and after follow-up (week 12)
  Six-minute walking test performed on a 30m flat surface. Participants walk maximally for 6 minutes with standardized encouragement. Distance recorded to nearest meter.Physiological responses (HR, SpO₂, RPE monitored) Total distance walked (meters)
Handgrip Strength | At baseline (week 0) and after follow-up (week 12)
  3 trials per hand, 30s rest between trials. Instrument: Jamar Hydraulic Hand Dynamometer. Highest value (kg)
Lower-limb muscle strength | At baseline (week 0) and after follow-up (week 12)
  Five-time sit to stand: Time to rise and sit from chair five times. Best time (seconds) of three trials with 30s rest.
Mobility | At baseline (week 0) and after follow-up (week 12)
  Timed Up-and-Go Test (TUG): Time to rise from chair, walk 3m, turn, return, and sit.
  Best time (seconds) of two trials.
Ambulatory blood pressure monitoring (ABPM) | At baseline (week 0) and after follow-up (week 12)
  Ambulatory systolic and diastolic blood pressure monitoring (ABPM), in millimeters of mercury (mmHg), will be measured for 24 hours after the end of each visit (approximately 90 minutes after the end of the Tai Chi, moderate-intensity combined exercise and control interventions), after a brief bath and using an automatic equipment (CardioMapa™, Cardios Sistemas Comercial e Industrial Ltda., São Paulo, Brazil).
Ambulatory heart rate variability (HRV) | At baseline (week 0) and after follow-up (week 12)
  Ambulatory systolic and diastolic blood pressure monitoring (ABPM), in millimeters of mercury (mmHg), will be measured for 24 hours after the end of each visit (approximately 90 minutes after the end of the Tai Chi, moderate-intensity combined exercise and control interventions), after a brief bath and using an automatic equipment (CardioMapa™, Cardios Sistemas Comercial e Industrial Ltda., São Paulo, Brazil).

OTHER OUTCOMES:
World Health Organization Quality of Life abbreviated (WHOQOL-BREF) scale | At baseline (week 0) and after follow-up (week 12)
  Change in health-related quality of life domains measured by the World Health Organization Quality of Life - Abbreviated Version (WHOQOL-BREF) scale (score range: 0-100), where higher scores indicate better quality of life.
World Health Organization Quality of Life Older Adults (WHOQOL-OLD) scale | At baseline (week 0) and after follow-up (week 12)
  Change in health-related quality of life domains measured by the World Health Organization Quality of Life - Older Adults (WHOQOL-OLD) scale (score range: 24-120), where higher scores indicate better quality of life.
Resting heart rate | Base line:Day 0 (before starting Tai Chi/MICE/CON) and post-intervention (Week 12)
  Heart rate will be measured using a digital telemetry system (Polar H10™, Polar Electro Inc, Kempele, Finland) in beats per minute (bpm)

IPD SHARING:
Plan to Share IPD: Yes
Participants who are interested in participating will provide an anamnesis to the investigator. The investigator will evaluate the IDP eligibility or non-eligibility criteria. Each qualified participant will get a document that includes the research protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code information. Thus, scientists will do cardiopulmonary activity tests to assess if IDP will be able to study the program
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be analysed after completing all 3 interventions (12week).
Access Criteria: Informed Consent Form described and signed. DP will received Informed Consent Form informing the objectives, study deling, interventions, analyses, risks and benefits. Participation in this study will be voluntary and confidential after signing of an informed consent
URL: https://plataformabrasil.saude.gov.br/